CLINICAL TRIAL: NCT06963346
Title: HERO Trial: Phase I Study Investigating Intravesical HDAC Inhibition to Improve Response to Immuno-Oncology Agents in Localized Bladder Cancer
Brief Title: Study Investigating Intravesical HDAC Inhibition to Improve Response to Immuno-Oncology Agents
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: H. Lee Moffitt Cancer Center and Research Institute (Other)
Collaborators: AstraZeneca (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: MCC-22623; ESR 23-22189 (Other: AstraZeneca)
Record Dates: First submitted 2025-04-29; First posted 2025-05-09 (Actual); Last update posted 2025-12-03 (Actual); Status verified 2025-12

CONDITIONS: Bladder Cancer
MeSH Terms: conditions — Urinary Bladder Neoplasms | interventions — romidepsin; durvalumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Dose Level 1 (Experimental): Romidepsin Level 1: 0.2 ng/ml on C1D1.
  Durvalumab: The recommended fixed dose of durvalumab is 1500 mg every 4 weeks and will be given on C1D1 and C2D1.
  Interventions: Drug: Romidepsin; Drug: Durvalumab
- Dose Level 2 (Experimental): Romidepsin Level 2: 0.4 ng/ml on C1D1.
  Durvalumab: The recommended fixed dose of durvalumab is 1500 mg every 4 weeks and will be given on C1D1 and C2D1.
  Interventions: Drug: Romidepsin; Drug: Durvalumab
- Dose Level 3 (Experimental): Romidepsin Level 3: 2.0 ng/m on C1D1.
  Durvalumab: The recommended fixed dose of durvalumab is 1500 mg every 4 weeks and will be given on C1D1 and C2D1.
  Interventions: Drug: Romidepsin; Drug: Durvalumab

INTERVENTIONS:
Drug: Romidepsin — Administered as intravesical treatment.
Drug: Durvalumab — Administered as intravenous treatment.

SUMMARY:
In this study, we aim to evaluate the safety and efficacy of neoadjuvant combination using intravesical romidepsin and durvalumab in cisplatin-ineligible patients with muscle invasive bladder cancer (MIBC).

ELIGIBILITY:
Inclusion Criteria:

* Patients must have histologically confirmed MIBC (T2-T4a, N0, M0 per American Joint Commission on Cancer [AJCC]) pure or mixed histology urothelial carcinoma.
* Patients must be ineligible for cisplatin-based chemotherapy due to any of the following: Creatinine clearance (CrCl) < 60 mL/min by the Cockcroft-Gault formula; Hearing impaired ≥ Grade 2 by CTCAE criteria; Neuropathy ≥ Grade 2 by CTCAE criteria; Heart failure NYHA ≥ III; ECOG ≥ 2.
* Patients must be medically fit for TURBT and radical cystectomy (RC
* Age ≥ 18 years
* Body weight >30 kg
* Ability to understand and willingness to sign IRB-approved informed consent.
* Willing to provide tumor tissue, blood, and urine samples for research.
* ECOG performance status 0 or 1 (Karnofsky ≥80%).
* Human immunodeficiency virus (HIV)-infected patients on effective anti-retroviral therapy with undetectable viral load within 6 months are eligible for this trial.
* For patients with evidence of chronic hepatitis B virus (HBV) infection, the HBV viral load must be undetectable on suppressive therapy, if indicated.
* Patients with a history of hepatitis C virus (HCV) infection must have been treated and cured. For patients with HCV infection who are currently on treatment, they are eligible if they have an undetectable HCV viral load.
* Participants must have adequate organ and marrow function as defined below: Hemoglobin ≥ 9.0 g/dL; Absolute neutrophil count (ANC) ≥ 1500/mcL; Platelet count ≥100,000/mcL; Serum bilirubin ≤1.5 x institutional upper limit of normal (ULN); total bilirubin must be < 3 x ULN for patients with Gilberts syndrome; AST (SGOT)/ALT (SGPT) ≤2.5 x institutional upper limit of normal; Measured creatinine CL >40 mL/min or Calculated creatinine CL>40 mL/min by the Cockcroft-Gault formula or by 24-hour urine collection for determination of creatinine clearance.
* Evidence of post-menopausal status or negative urinary or serum pregnancy test for female pre-menopausal patients.
* Non-sterile males must be willing to use a highly effective method of birth control for the duration of the study and for ≥120 days after the last dose of durvalumab.
* Patient is willing and able to comply with the protocol for the duration of the study including undergoing treatment and scheduled visits and examinations including follow up.
* Patient must have a life expectancy of at least 12 weeks

Exclusion Criteria:

* Patients with active or prior documented autoimmune disease within the past 2 years prior to Screening or other immunosuppressive agent within 14 days of study treatment. NOTE: Patients with well controlled type 1 diabetes mellitus, vitiligo, Graves' disease, Hashimoto's disease, eczema, lichen simplex chronicus, or psoriasis not requiring systemic treatment (within the past 2 years prior to Screening) are not excluded.
* Patients who have concurrent upper urinary tract (i.e. ureter, renal pelvis) invasive urothelial carcinoma. Patients with history of non-invasive (Ta, T1, Tis) upper tract urothelial carcinoma that has been definitively treated with at least one post-treatment disease assessment (i.e. cytology, biopsy, imaging) that demonstrates no evidence of residual disease are eligible.
* Patients who have another malignancy that could interfere with the evaluation of safety or efficacy of the study drugs. Patients with a prior malignancy will be allowed without Principal Investigator approval in the following circumstances: Not currently active and diagnosed at least 5 years prior to the date of registration; Non-invasive diseases such as low risk cervical cancer or any cancer in situ; Localized (early stage) cancer treated with curative intent (without evidence of recurrence and intent for further therapy), and in which no chemotherapy was indicated (e.g. low/intermediate risk prostate cancer, etc.). Patients with other malignancies not meeting these criteria must be discussed prior to registration.
* Patients who have received any prior immune checkpoint inhibitor (i.e. anti-KIR, anti-PD-1, anti- PD-L1, (including durvalumab) anti-CTLA4 or other).
* Patients who have undergone major surgery (e.g. intra-thoracic, intra-abdominal or intra-pelvic), open biopsy or significant traumatic injury or specific anti-cancer treatment ≤ 4 weeks prior to starting study drug, or patients who have had placement of vascular access device ≤ 1 week prior to starting study drug, or who have not recovered from side effects of such procedure or injury.
* Patients who have clinically significant cardiac diseases deemed not fit for radical cystectomy, including any of the following: History or presence of serious uncontrolled ventricular arrhythmias; Clinically significant resting bradycardia; Any of the following within 3 months prior to starting study drug: severe/unstable angina, Congestive Heart Failure (CHF), Cerebrovascular Accident (CVA), Transient Ischemic Attack (TIA); Uncontrolled hypertension defined by a SBP ≥ 180 mm Hg and/or DBP ≥ 100 mm Hg, with or without anti-hypertensive medication(s).
* Patients who have history of chronic active liver disease or evidence of acute or chronic Hepatitis B Virus (HBV) or Hepatitis C (HCV).
* Patients who have known diagnosis of human immunodeficiency virus (HIV) infection. Testing is not required in absence of clinical suspicion.
* Patients who have known diagnosis of any condition (e.g. post-hematopoietic or solid organ transplant, pneumonitis, inflammatory bowel disease, etc.) that requires chronic immunosuppressive therapy which cannot be stopped for the duration of the clinical trial. Usage of non-steroidal anti-inflammatory medications (NSAIDS) for the treatment of osteoarthritis and uric acid synthesis inhibitors for the treatment of gout are permitted.
* Patients with any serious and/or uncontrolled concurrent medical conditions.
* Patients who have used any live viral vaccine for prevention of infectious diseases within 4 weeks prior to study drug(s). Examples of live vaccines include, but are not limited to, the following: measles, mumps, rubella, varicella/zoster (chicken pox), yellow fever, rabies, BCG, and typhoid vaccine. Seasonal influenza vaccines for injection are generally killed virus vaccines and are allowed; however, intranasal influenza vaccines (e.g., FluMist®) are live attenuated vaccines and are not allowed. COVID vaccination is allowed.
* Patients unwilling or unable to comply with the protocol.
* Patients with a known allergy to any of the study medications, their analogues, or excipients in the various formulations of any agent.
* Patients who participate in any other therapeutic clinical trials, including those with other investigational agents not included in this trial throughout the duration of this study.
* Patients receiving any medications or substances that are strong inhibitors or inducers of CYP3A are ineligible. Because the lists of these agents are constantly changing, it is important to regularly consult a frequently-updated medical reference.
* Patients with local symptoms from bladder cancer, (e.g. gross hematuria, dysuria, etc.) who are deemed to be unable to complete the treatment protocol per PI.
* Any concurrent chemotherapy, IP, biologic, or hormonal therapy for cancer treatment. Concurrent use of hormonal therapy for non-cancer-related conditions (e.g., hormone replacement therapy) is acceptable.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Estimated)
Dates: Start 2025-06-24 (Actual); Primary Completion 2028-04 (Estimated); Study Completion 2028-04 (Estimated)

PRIMARY OUTCOMES:
Romidepsin Maximum Tolerated Dose (MTD) | Up to 28 days
  The MTD will be estimated using isotonic regression based on observed DLT from all DLT-evaluable patients.

SECONDARY OUTCOMES:
Pathological Response | Up to 1 year
  Pathologic response is defined as <pT2N0 disease at the time of RC (e.g. pT0N0, pT1N0, pTaN0, or pTisN0).
Pathologic complete response (pCR) | Up to 1 year
  Pathologic complete response (pCR) is defined as achievement of pT0N0 disease at RC.
Relapse-free survival (RFS) | Up to 1 year
  Relapse-free survival (RFS) is defined as the duration of time from time of RC to time of documented disease relapse or recurrence after RC, or death from any cause.

CONTACTS AND LOCATIONS:
Overall Officials: Jingsong Zhang, MD, PhD, Principal Investigator — Moffitt Cancer Center
Locations (1):
- Moffitt Cancer Center, Tampa, Florida, United States